CLINICAL TRIAL: NCT02368210
Title: A Multicenter, Randomized, Double-Blind, Parallel Group Comparison of 122-0551 Foam Versus Vehicle Foam in Subjects With Plaque Psoriasis (Study 306)
Brief Title: A Comparison of 122-0551 Foam Versus Vehicle Foam in Subjects With Plaque Psoriasis (Study 306)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 122-0551-306
Record Dates: First submitted 2015-02-13; First posted 2015-02-23 (Estimated); Results first posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-10

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 122-0551 Foam (Experimental): 122-0511 Foam, topically applied twice daily
  Interventions: Drug: 122-0551 Foam
- Vehicle Foam (Placebo Comparator): Vehicle Foam, topically applied twice daily
  Interventions: Drug: Vehicle Foam

INTERVENTIONS:
Drug: 122-0551 Foam — Topical Foam
  Arms: 122-0551 Foam
Drug: Vehicle Foam — Topical Foam
  Arms: Vehicle Foam

SUMMARY:
This Phase 3 study (Study 306) has been designed to determine and compare the efficacy and safety of 122-0551 Foam and Vehicle Foam applied twice daily for two weeks in subjects with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a clinical diagnosis of stable plaque psoriasis involving a minimum of 2% and no more than 12% affected body surface area.
* Subject has an Investigator's Global Assessment (IGA) score of at least three (moderate) at study start.
* If subject is a woman of childbearing potential, she must have a negative urine pregnancy test and agree to use an effective form of birth control for the duration of the study.

Exclusion Criteria:

* Subject has spontaneously improving or rapidly deteriorating plaque psoriasis.
* Subject has guttate, pustular, erythrodermic or other non-plaque forms of psoriasis.
* Subject has a physical condition which, in the investigator's opinion, might impair evaluation of plaque psoriasis, or which exposes the subject to an unacceptable risk by study participation.
* Subject has used any phototherapy (including laser), photo-chemotherapy or other forms of photo based therapy for the treatment of their psoriasis within 30 days prior to study start.
* Subject has used any systemic methotrexate, retinoids, systemic corticosteroids [including intralesional, intra-articular, and intramuscular corticosteroids], cyclosporine or analogous products within 90 days prior to study start.
* Subject has used any systemic biologic therapy (i.e., FDA-approved or experimental therapy) within five half-lives of the biologic prior to study start.
* Subject had prolonged exposure to natural or artificial sources of ultraviolet radiation within 30 days prior to study start or is intending to have such exposure during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Andrasfay, Study Director — Therapeutics, Inc.
Locations (8):
- United States (8):
  - Center for Dermatology Clinical Research, Fremont, California
  - International Dermatology Research, Inc., Miami, Florida
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Dermatology Associates of Knoxville, Knoxville, Tennessee
  - The Center for Skin Research, Houston, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

REFERENCES:
- [Derived] Bhatia N, Stein Gold L, Kircik LH, Schreiber R. Two Multicenter, Randomized, Double-Blind, Parallel Group Comparison Studies of a Novel Foam Formulation of Halobetasol Propionate, 0.05% vs Its Vehicle in Adult Subjects With Plaque Psoriasis. J Drugs Dermatol. 2019 Aug 1;18(8):790-796. PMID 31424709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: January 2015 to June 2015
  The location of clinical sites included dermatology clinics and clinical research centers.
Pre-assignment Details: All subjects who met the entry criteria were randomized and enrolled into the study.
Period: Overall Study
Arm/Group | 122-0551 Foam | Vehicle Foam
Started | 75 | 76
Completed | 74 | 75
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographics data is based on the Intent-To-Treat (ITT) population, defined as all enrolled subjects in the study who were randomized and dispensed the test article.
Groups:
- Total: Total of all reporting groups
Arm/Group | 122-0551 Foam | Vehicle Foam | Total
Number analyzed (Participants) | 75 | 76 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (14.22) | 55.1 (13.86) | 54.5 (14.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 49
  Male | 48 | 54 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 22 | 43
  Not Hispanic or Latino | 54 | 54 | 108
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 6 | 15
  White | 63 | 68 | 131
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75 | 76 | 151

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Rated a "Treatment Success" Based on the Investigator's Global Assessment (IGA)
Description: The IGA score is a static evaluation of the overall or "average" degree of severity of a subject's disease, taking into account all of the subject's psoriatic lesions. "Treatment success" is defined as a score of 0 or 1 representing "cleared" or "almost cleared" at Day 15 with at least a two grade decrease in severity score relative to Baseline. IGA is measured on a 5-point scale, ranging from 0 (clear) to 4 (severe/very severe).
Time Frame: Day 15
Population: Analysis shown is based on the ITT population, defined as all enrolled participants who were randomized and applied at least one dose of the test article.
Measure: Number; unit: percentage of participants
Arm/Group | 122-0551 Foam | Vehicle Foam
Number analyzed (Participants) | 75 | 76
percentage of participants | 25.3 | 3.9
Statistical Analysis 1: Comparison: 122-0551 Foam vs Vehicle Foam; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Treatment groups were compared with respect to the proportions of subjects with "treatment success" at Day 15 using the Cochran-Mantel-Haenszel (CMH) test stratified by analysis center; Missing data was imputed as treatment failure

2. Secondary Outcome: Percentage of Subjects Rated a "Treatment Success" for Each of the Clinical Signs of Psoriasis (Scaling, Erythema and Plaque Elevation)
Description: A static assessment of the overall or "average" degree of severity of each of three key characteristics present within all of the subject's psoriatic lesions. "Treatment success" is defined as a score of 0 or 1 representing "cleared" or "almost cleared" at Day 15 with at least a two grade decrease in severity score relative to Baseline. Each clinical sign of psoriasis is measured on a 5-point scale, ranging from 0 (clear) to 4 (severe/very severe).
Time Frame: Day 15
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 122-0551 Foam | Vehicle Foam
Number analyzed (Participants) | 75 | 76
percentage of participants
  Scaling | 28.0 | 5.3
  Erythema | 21.3 | 2.6
  Plaque Elevation | 26.7 | 3.9
Statistical Analysis 1: Comparison: 122-0551 Foam vs Vehicle Foam; Treatment groups were compared with respect to each of the clinical signs of psoriasis (scaling, erythema and plaque elevation); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The pre-specified threshold for statistical significance was ≤0.05. The reported P-Value applies to the clinical sign of psoriasis: Scaling; Missing data was imputed as treatment failure
Statistical Analysis 2: Comparison: 122-0551 Foam vs Vehicle Foam; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The pre-specified threshold for statistical significance was ≤0.05. The reported P-Value applies to the clinical sign of psoriasis: erythema; Missing data was imputed as treatment failure
Statistical Analysis 3: Comparison: 122-0551 Foam vs Vehicle Foam; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — The pre-specified threshold for statistical significance was ≤0.05. The reported P-Value applies to the clinical sign of psoriasis: Plaque Elevation; Missing data was imputed as treatment failure

3. Other Pre Specified Outcome: Percentage of Subjects With IGA "Treatment Success"
Description: "Treatment success" and IGA as defined in the primary outcome measure. "Treatment success" is defined as a score of 0 or 1 representing "cleared" or "almost cleared" at Day 15 with at least a two grade decrease in severity score relative to Baseline. IGA is measured on a 5-point scale, ranging from 0 (clear) to 4 (severe/very severe).
Time Frame: Day 8
Population: Analysis shown is based on the Intent-to-Treat (ITT) population and observed results.
Measure: Number; unit: percentage of participants
Arm/Group | 122-0551 Foam | Vehicle Foam
Number analyzed (Participants) | 75 | 76
percentage of participants | 8.1 | 2.6

4. Other Pre Specified Outcome: Percentage of Subjects Rated a "Treatment Success" for Each of the Clinical Signs of Psoriasis (Scaling, Erythema and Plaque Elevation)
Description: "Treatment success" and clinical signs as defined in the secondary outcome measure. "Treatment success" is defined as a score of 0 or 1 representing "cleared" or "almost cleared" at Day 15 with at least a two grade decrease in severity score relative to Baseline. Each clinical sign of psoriasis is measured on a 5-point scale, ranging from 0 (clear) to 4 (severe/very severe).
Time Frame: Day 8
Population: Analysis shown is based on the Intent-to-Treat (ITT) population and observed results.
Measure: Number; unit: percentage of participants
Arm/Group | 122-0551 Foam | Vehicle Foam
Number analyzed (Participants) | 75 | 76
percentage of participants
  Scaling | 12.2 | 3.9
  Erythema | 10.8 | 1.3
  Plaque Elevation | 10.8 | 3.9

5. Other Pre Specified Outcome: Change From Baseline in Pruritus Score
Description: Pruritus scale will be used to assess the subjective and multidimensional experience of the subject's pruritus (itching) during the previous two weeks at Baseline and Day 15. Possible scores range from 5 (no pruritus) to 25 (most severe pruritus).
Time Frame: Baseline and Day 15
Population: Analysis shown is based on the Intent-to-Treat (ITT) population and observed results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 122-0551 Foam | Vehicle Foam
Number analyzed (Participants) | 75 | 76
units on a scale | -4.4 (4.03) | -2.0 (3.19)

6. Other Pre Specified Outcome: Change in Percent Body Surface Area (BSA) With Active Psoriasis
Description: The investigator will use the assumption that 1% BSA is approximately equal to the surface area of the subject's palm and fingers, with the fingers extended yet grouped together, creating a flat oval-like surface area.
Time Frame: Baseline and Day 15
Population: Analysis shown is based on the Intent-to-Treat (ITT) population and observed results.
Measure: Mean (Standard Deviation); unit: Change in percent BSA
Arm/Group | 122-0551 Foam | Vehicle Foam
Number analyzed (Participants) | 75 | 76
Change in percent BSA
  Baseline % BSA | 5.7 (3.09) | 5.7 (3.22)
  Change in % BSA at Day 15 | -0.9 (1.56) | -0.2 (0.69)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from study Day 1 (enrollment/first dose) to study completion (Day 15) or participant termination. AEs that continued beyond completion/termination were followed until resolution or stabilization.
Description: The safety population included all participants enrolled in the study who were dispensed and applied the test article at least once; because the first dose of the test article was applied at the study site (Day 1), all participants (N=151) were included in the safety population. Subjects reporting a particular AE more than once are counted only once for that AE.
Arm/Group | 122-0551 Foam | Vehicle Foam
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/76
Other Adverse Events (participants affected / at risk) | 5/75 | 3/76
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 122-0551 Foam (N=75) | Vehicle Foam (N=76)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site pain (General disorders) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Laceration (Infections and infestations) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 12 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review thirty days prior to public disclosure. The PI may not disclose previously undisclosed confidential information other than study results.